CLINICAL TRIAL: NCT05203068
Title: Evaluation of the Specificity of Intradermal Test With Recombinant Tuberculosis Allergen in BCG Vaccinated Healthy Volunteers
Brief Title: Specificity Trial of the Recombinant Tuberculosis Allergen in BCG Vaccinated Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Medical Research Center of Phthisiopulmonology and Infectious Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 102/1
Record Dates: First submitted 2022-01-09; First posted 2022-01-24 (Actual); Results first posted 2023-08-25 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2022-10

CONDITIONS: Tuberculosis
Keywords: Tuberculosis; TB diagnosis; Tuberculosis skin test; CFP10; ESAT6
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Recombinant tuberculosis allergen (CFP10-ESAT6) (Experimental): RTA (CFP10-ESAT6) 0.2 µg/0.1 mL RTA given intradermally on the middle of the forearm
  Interventions: Diagnostic Test: Recombinant tuberculosis allergen (RTA)

INTERVENTIONS:
Diagnostic Test: Recombinant tuberculosis allergen (RTA) — Single intradermal application of 0.2 µg/0.1 mL RTA (CFP10-ESAT6) in the middle of the forearm
  Other Names: Diaskintest

SUMMARY:
The aim of this study is to test the recombinant tuberculosis skin test in the previously BCG vaccinated healthy adults with low risk of TB development, to determine the test specificity.

DETAILED DESCRIPTION:
Recombinant tuberculosis allergen (RTA) is a recombinant fusion protein CFP10-ESAT6 produced by the prokaryotic cell line. The test is widely used in Russian Federation and CIS countries for the latent TB diagnosis in adults and children over 8 years old. The current clinical study is a prospective, multicenter, open-label study in the cohort of healthy adults, not classified as at risk of tuberculosis, with no clinical symptoms of the disease, with a negative T-SPOT.TB test results, to evaluate the specificity of the RTA test in 72 hours following administration of the product at a dose of 0.2 μg/0.1 mL.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent for the participation in the study.
2. Age 18 to 30 years
3. A history of BCG vaccination (confirmed by medical documentation and/or the presence of BCG scar)
4. Healthy individual according to physical examination and medical records at screening.
5. Willingness to cooperate and follow the recommendations of the Investigator in accordance with the Protocol.

Exclusion Criteria:

1. A history of tuberculosis or close contact with a patient with active tuberculosis for 5 years prior to the enrollment in the study.
2. Positive T-SPOT.TB test at the enrollment in the study
3. Treatment with drugs affecting immune system within 3 months prior to the enrollment in the study
4. Vaccination against any infections <1.5 months prior to the enrollment in the study
5. Vaccination with BCG <6 months prior to the enrollment in the study.
6. The Mantoux test with 2 TU and/or the test with the recombinant tuberculosis allergen was performed less than 6 months prior to the enrollment in the study.
7. Congenital or acquired immunodeficiency.
8. Active disease of the immune system
9. HIV infection.
10. The current condition of the skin interferes with the conduct and reading of skin tests (trauma, skin diseases).
11. A disease in which blood sampling poses a risk to the volunteer (hemophilia, other bleeding disorders) or obstructed venous access.
12. The volunteer currently participates in another clinical study or has participated in another clinical study within 3 months prior to the enrollment in the study.
13. Previous participation in clinical studies of ESAT-6 and/or CFP-10 antigens.
14. Pregnancy, lactation, pregnancy planning.
15. The reluctance of a female person to use effective barrier (including spermicidal gel), hormonal or intrauterine contraceptives during the study.
16. History of alcohol, drug, benzodiazepine, or other substance abuse within the 12 months prior to the enrollment in the study.
17. Use of alcoholic beverages within 24 hours prior to the visit.
18. A condition or disease that, in the opinion of the Investigator, is inappropriate for participation in the study.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2021-11-24 (Actual); Primary Completion 2022-01-18 (Actual); Study Completion 2022-01-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aleksey V. Kazakov, MD, Principal Investigator — National Medical Research Center of Phthisiopulmonology and Infectious Diseases; Anastasia G. Samoylova, MD, Study Chair — National Medical Research Center of Phthisiopulmonologyand Infectious Diseases; Valentina A. Aksyonova, Prof., Study Chair — National Medical Research Center of Phtisiopulmonology and Infectious Diseases
Locations (1):
- National Medical Research Center of Phthisiopulmonology and Infectious Diseases, Moscow, Russia

REFERENCES:
- [Derived] Vasilyeva IA, Aksenova VA, Kazakov AV, Kiseleva YY, Maryandyshev AO, Dolzhenko EN, Abramchenko AV, Klevno NI, Glebov KA, Panova AE, Petrova LY, Sheikis EG, Seregina IV, Nikishova EI, Doktorova NP, Samoilova AG. Evaluation of the specificity of an intradermal test with recombinant tuberculosis allergen in Bacillus Calmette-Guerin-vaccinated healthy volunteers. Front Med (Lausanne). 2023 Mar 1;10:1042461. doi: 10.3389/fmed.2023.1042461. eCollection 2023. PMID 36936243

RESULTS

PARTICIPANT FLOW:
Period: RTA Result Assessment, 72 Hours
Arm/Group | Recombinant Tuberculosis Allergen (CFP10-ESAT6)
Started | 150
Completed | 150
Not Completed | 0
Period: RTA Safety Assessment, 28 Days
Arm/Group | Recombinant Tuberculosis Allergen (CFP10-ESAT6)
Started | 150
Completed | 150
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 150 healthy adult subjects
Arm/Group | Recombinant Tuberculosis Allergen (CFP10-ESAT6)
Number analyzed (Participants) | 150
Age, Continuous [Mean (Full Range); unit: years] | 21.5 [20 to 22]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 122
  Male | 28
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Russia | 150
Body weight [Mean (Full Range); unit: kilograms] | 60 [55 to 69]
BCG-vaccination history [Count of Participants; unit: Participants] | 150
Having allergic diseases in the past [Count of Participants; unit: Participants] | 148
Having chronic diseases [Count of Participants; unit: Participants] | 8
COVID-19 vaccinated [Count of Participants; unit: Participants] | 145

OUTCOME MEASURES:

1. Primary Outcome: Number of the Volunteers With the True Negative RTA Result
Description: Absolute number and percentage of the volunteers with negative and positive test results with RTA based on the results of the assessment of the infiltrate 72 hours after the test application
Time Frame: hour 72
Measure: Count of Participants; unit: Participants
Arm/Group | Recombinant Tuberculosis Allergen (CFP10-ESAT6)
Number analyzed (Participants) | 150
Participants
  Count RTA negative | 145
  Count RTA positive | 5

2. Secondary Outcome: Number of Subjects With Local Adverse Reactions Within 72 Hours Following the Intradermal Test Application
Description: To assess the number of subjects who developed the injection site adverse reaction (redness, swelling etc) within 72 hours after RTA test application
Time Frame: hour 72
Measure: Count of Participants; unit: Participants
Arm/Group | Recombinant Tuberculosis Allergen (CFP10-ESAT6)
Number analyzed (Participants) | 150
Participants | 0

3. Secondary Outcome: Number of Participants With General and Local Adverse Reactions Within 28 Days After Administration of RTA
Description: To assess the number of subjects who developed the general adverse reaction (e.g. infections, fever, headache, weakness etc) based on the subjects complaints and physical examination, and local injection site reaction (redness, swelling etc) up to 28 days after intradermal RTA application.
Time Frame: Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Recombinant Tuberculosis Allergen (CFP10-ESAT6)
Number analyzed (Participants) | 150
Participants
  Number of participants developed general adverse reaction in 28 days after RTA application | 1
  Number of participants developed local adverse reactions in 28 days after RTA application | 0
  Number of participants without adverse reactions in 28 days after RTA application | 149

ADVERSE EVENTS:
Time Frame: 28 days
Arm/Group | Recombinant Tuberculosis Allergen (CFP10-ESAT6)
All-Cause Mortality (participants affected / at risk) | 0/150
Serious Adverse Events (participants affected / at risk) | 0/150
Other Adverse Events (participants affected / at risk) | 1/150
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Recombinant Tuberculosis Allergen (CFP10-ESAT6) (N=150)
Respiratory tract infection (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-22): https://cdn.clinicaltrials.gov/large-docs/68/NCT05203068/Prot_SAP_000.pdf